CLINICAL TRIAL: NCT03950167
Title: Gallbladder Functions & Serum Cholecystokinin Levels in Pregnant Women Diagnosed With Hyperemesis Gravidarum
Brief Title: Gallbladder Functions & Serum Cholecystokinin Levels in Women Diagnosed With Hyperemesis Gravidarum
Status: Completed | Type: Observational
Sponsor: Müge Keskin (Other)
Responsible Party: Sponsor-Investigator, Müge Keskin, Principal investigator, Ufuk University
Organization: Ufuk University (Other)
Other Study IDs: 20190328
Record Dates: First submitted 2019-04-30; First posted 2019-05-15 (Actual); Results first posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Hyperemesis Gravidarum; Pregnancy Related
Keywords: gallbladder functions; cholecystokinin; hyperemesis gravidarum
MeSH Terms: conditions — Hyperemesis Gravidarum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hyperemesis gravidarum: pregnant women before 14 weeks of pregnancy diagnosed with hyperemesis gravidarum will be assessed in terms of gallbladder functions and serum cholecystokinin levels after a fatty meal.
- Healthy pregnant women: Healthy pregnant women before 14 weeks of pregnancy without hyperemesis gravidarum will be assessed in terms of gallbladder functions and serum cholecystokinin levels after a fatty meal.

SUMMARY:
This study evaluates the gallbladder functions and serum cholecystokinin levels in pregnant women diagnosed with hyperemesis gravidarum. Half of the participants are healthy pregnant women and half of the participants are pregnant women diagnosed with hyperemesis gravidarum. Two groups will be compared by means of gallbladder functions and serum cholecystokinin levels.

DETAILED DESCRIPTION:
Previously gallbladder functions have been observed in human with gallbladder disease. However it has never been evaluated whether there is any difference in gallbladder functions between healthy pregnant women and pregnant women diagnosed with hyperemesis gravidarum. Moreover correlation between hyperemesis gravidarum symptom scores and gallbladder functions has never been assessed. There is also few data comparing serum cholecystokinin levels between healthy pregnant women and those diagnosed with hyperemesis gravidarum. The investigators will measure serum cholecystokinin levels after a fatty meal (100 g chocolate) and compare two groups. In this study the investigators would like to evaluate gallbladder functions and serum cholecystokinin levels in women with hyperemesis gravidarum and compare these with healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* gestation week between 6 and 14 weeks,
* singleton pregnancy with a live embryo,
* healthy women without any medical disorders,

Exclusion Criteria

* any systemic disease,
* gallbladder disease
* any psychological disorder that can cause vomiting,
* multiple gestation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: healthy pregnant women and pregnant women diagnosed with hyperemesis gravidarum before 14 weeks of pregnancy
Sampling Method: Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muge Keskin, Principal Investigator — Ufuk University
Locations (1):
- Ufuk University Hospital, Ankara, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a prospective cohort study conducted in Ufuk University hospital, Ankara, Turkey (a tertiary center) between March 2019 and May 2020.
Pre-assignment Details: Excluded (n=275)
  * Not meeting inclusion criteria (n=163) Inclusion criteria were: gestation week between 6 and 14 weeks, singleton pregnancy with a live embryo, age range between 18 and 40 years, healthy women without any medical disorders, Women with any systemic disease, gallbladder disease or any psychological disorder that can cause vomiting, multiple gestation were excluded.
  * Declined to participate (n=112)
Period: Overall Study
Arm/Group | Hyperemesis Gravidarum | Healthy Pregnant Women
Started | 25 | 25
Completed | 24 | 22
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Population: PREGNANT WOMEN DİAGNOSED WITH HYPEREMESİS GRAVIDARUM AND HEALTHY PREGNANT WOMEN
Groups:
- Total: Total of all reporting groups
Arm/Group | Hyperemesis Gravidarum | Healthy Pregnant Women | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] — women aged between 18-40 were recruited
  years | 30.08 (4.03) | 30.91 (4.20) | 30.49 (2.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 46
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 24 | 22 | 46
Region of Enrollment [Number; unit: participants]
  Turkey | 24 | 22 | 46
age [Mean (Standard Deviation); unit: years] — Age, continuous
  years | 30.91 (4.2) | 30.08 (4.03) | 30.49 (4.11)
body mass index (BMI) [Mean (Standard Deviation); unit: kg/m²] — weight in kilograms divided by the square of height in meters
  kg/m² | 23.95 (3.53) | 24.55 (4.72) | 24.25 (4.125)
gravidity [Median (Inter-Quartile Range); unit: gravidity] — the number of times that a woman has been pregnant
  gravidity | 2 [1 to 2] | 2 [2 to 3] | 2 [1 to 3]
Gestational age [Median (Full Range); unit: weeks] — description of how far along the pregnancy is. It is measured in weeks
  weeks | 9.07 [6.14 to 13] | 8.92 [6.28 to 13.5] | 8.995 [6.21 to 13.25]
parity [Median (Inter-Quartile Range); unit: parity] — the number of times that a woman has given birth a fetus with a gestational age of 24 weeks or more
  parity | 1 [0 to 1] | 1 [0 to 1] | 1 [0 to 1]

OUTCOME MEASURES:

1. Primary Outcome: Blood Cholecystokinin (CCK) Levels
Description: a gut hormone released, its level can be measured in blood as fasting level and postprandial
Time Frame: Fasting (baseline) and postprandial (15 minutes after the test meal) CCK level
Measure: Mean (Standard Deviation); unit: picogram/mililiters (pg/ml)
Arm/Group | Hyperemesis Gravidarum | Healthy Pregnant Women
Number analyzed (Participants) | 24 | 22
picogram/mililiters (pg/ml)
  fasting CCK | 53.13 (25.3) | 54.55 (25.32)
  postprandial CCK | 73.61 (30.29) | 81.24 (29.89)
Statistical Analysis 1: Comparison: Hyperemesis Gravidarum vs Healthy Pregnant Women; Test type: Other; p = 0.05, t-test, 2 sided — A p value of <0.05 was accepted as significant in all statistical analyses; Mean Difference (Final Values) = 0.85 — p value demonstrated above is the calculated value. Fasting CCK level difference: hyperemesis group-control group
Statistical Analysis 2: Comparison: Hyperemesis Gravidarum vs Healthy Pregnant Women; Since this is the first study comparing both CCK levels and GB functions in patients diagnosed with hyperemesis gravidarum (HG) and healthy pregnant women, a power analysis was not feasible; Test type: Other; p = 0.05, t-test, 2 sided; Mean Difference (Net) = 0.68 — p value demonstrated above is the calculated value. Postprandial CCK level difference: hyperemesis group-control group

2. Primary Outcome: Gallbladder (GB) Wall Thickness
Description: GB wall thickening measured with abdominal ultrasound at fasting and postprandial
Time Frame: fasting and postprandial 45th minute
Measure: Mean (Standard Deviation); unit: milimeters (mm)
Arm/Group | Hyperemesis Gravidarum | Healthy Pregnant Women
Number analyzed (Participants) | 24 | 22
milimeters (mm)
  fasting GB wall thickness | 2.10 (0.57) | 2.11 (0.47)
  postprandial GB wall thickness | 2.51 (0.51) | 2.74 (0.76)
Statistical Analysis 1: Comparison: Hyperemesis Gravidarum vs Healthy Pregnant Women; Test type: Other; p = 0.05, t-test, 2 sided — A p value of <0.05 was accepted as significant in all statistical analyses; Mean Difference (Final Values) = 0.91 — p value demonstrated above is the calculated value. Fasting GB wall thickness: Hyperemesis group-control group
Statistical Analysis 2: Comparison: Hyperemesis Gravidarum vs Healthy Pregnant Women; Test type: Other; p = 0.05, t-test, 2 sided — A p value of <0.05 was accepted as significant in all statistical analyses; Mean Difference (Final Values) = 0.23 — p value demonstrated above is the calculated value. Postprandial GB wall thickness: hyperemesis group-control group

3. Primary Outcome: Gallbladder (GB) Volume
Description: volume of GB measured with abdominal ultrasound at fasting and postprandial
Time Frame: fasting and postprandial 45th minute
Measure: Mean (Standard Deviation); unit: mililiter (ml)
Arm/Group | Hyperemesis Gravidarum | Healthy Pregnant Women
Number analyzed (Participants) | 24 | 22
mililiter (ml)
  fasting GB volume | 36.9 (13.8) | 33.69 (12.54)
  postprandial GB volume | 17.29 (8.14) | 18.33 (6.98)
Statistical Analysis 1: Comparison: Hyperemesis Gravidarum vs Healthy Pregnant Women; Test type: Other; p = 0.05, t-test, 2 sided — A p value of <0.05 was accepted as significant in all statistical analyses; Mean Difference (Final Values) = 0.41 — p value demonstrated above is the calculated value. Fasting GB volume: hyperemesis group-control group
Statistical Analysis 2: Comparison: Hyperemesis Gravidarum vs Healthy Pregnant Women; Test type: Other; p = 0.05, t-test, 2 sided — A p value of <0.05 was accepted as significant in all statistical analyses; Mean Difference (Final Values) = 0.71 — p value demonstrated above is the calculated value. Postprandial GB volume: hyperemesis group-control group

4. Primary Outcome: Gallbladder (GB) Ejection Fraction
Description: GB ejection fraction measures how much bile gallbladder releases at one time, expressed as percentage
Time Frame: The fasting and postprandial 45th minute
Measure: Mean (Standard Deviation); unit: Percantage (%)
Arm/Group | Hyperemesis Gravidarum | Healthy Pregnant Women
Number analyzed (Participants) | 24 | 22
Percantage (%) | 52.06 (19.45) | 45.46 (16.59)
Statistical Analysis 1: Comparison: Hyperemesis Gravidarum vs Healthy Pregnant Women; Test type: Other; p = 0.05, t-test, 2 sided — A p value of <0.05 was accepted as significant in all statistical analyses; Mean Difference (Final Values) = 0.22 — p value demonstrated above is the calculated value. Fasting GB ejection fraction: hyperemesis group-control group
Statistical Analysis 2: Comparison: Hyperemesis Gravidarum vs Healthy Pregnant Women; Test type: Other; p = 0.05, t-test, 2 sided — A p value of <0.05 was accepted as significant in all statistical analyses; Mean Difference (Final Values) = 0.63 — p value demonstrated above is the calculated value. Postprandial GB ejection fraction: hyperemesis group-control group

ADVERSE EVENTS:
Time Frame: 1 year 6 months
Description: a fatty test meal (100 g milk chocolate) was given to all participants for the evaluation of postprandial cholecystokinin levels and gallbladder parameters including volume and gallbladder wall thickness. Nausea and vomiting are the possible adverse events that may have been observed.
Arm/Group | Hyperemesis Gravidarum | Healthy Pregnant Women
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/22
Other Adverse Events (participants affected / at risk) | 0/24 | 0/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hyperemesis Gravidarum (N=24) | Healthy Pregnant Women (N=22)
Nausea and vomitting (Gastrointestinal disorders) | 0 | 0 — Nausea and vomiting after fatty meal (100 g milk chocolate)

LIMITATIONS AND CAVEATS:
Lack of power analysis and inclusion of few patients after assessing eligibility for the study are the limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT03950167/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT03950167/ICF_001.pdf